CLINICAL TRIAL: NCT00248664
Title: A Case Control Study of Interstitial Cystitis
Brief Title: Events Preceding Interstitial Cystitis (EPIC)
Acronym: EPIC
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: DK64880 (completed)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-03

CONDITIONS: Cystitis, Interstitial
Keywords: Cystitis, Interstitial; Case-Control Studies; Risk Factors
MeSH Terms: conditions — Cystitis, Interstitial

SUMMARY:
EPIC is a case/control study that seeks to identify the risk factors for interstitial cystitis by comparing the experiences and medical histories of 400 women who recently developed IC with 400 similar people who do not have the disease.

DETAILED DESCRIPTION:
This project is a systematic, national study of incident IC cases and controls matched by age and gender. By telephone interview and medical record review, we compare exposures of cases and controls seeking significant differences which may be risk factors for IC. This cohort of incident IC cases will initiate a natural history study of the disease.

Specific Aim 1. To test the hypothesis that certain features that precede onset of IC symptoms, e.g., bacterial cystitis, distinguish IC cases from controls matched for age and gender, and may be risk factors for the disease.

Specific Aim 2. To test the hypotheses that patients with IC have higher prevalences of certain non bladder syndromes, e.g., irritable bowel syndrome, than do controls matched for age and gender.

Specific Aim 3. To test the hypothesis that urine APF, HB EGF, and/or EGF are sensitive and specific diagnostic markers for IC in patients with symptoms of ÿ12 months.

Specific Aim 4. To test the hypotheses that, in an incident cohort, patients with IC have remissions and that certain clinical features, e.g., bacterial cystitis at disease onset, are prognostic factors for remissions.

ELIGIBILITY:
Inclusion Criteria: Female Adults(18 and over) who have had symotoms of IC for 12 months or fewer

-

Exclusion Criteria: Males,children, those who do not have symptoms of IC or those who have had symtoms for greater than 12 months.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2004-03; Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W Warren, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States